CLINICAL TRIAL: NCT02796118
Title: ASP2151 Phase 1 Study - Multiple Oral Dosing Study in Healthy Non-elderly Male and Elderly Male Japanese Subjects-
Brief Title: Study to Evaluate the Safety and Pharmacokinetics of ASP2151 in Healthy Non-elderly and Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15L-CL-003
Record Dates: First submitted 2016-06-07; First posted 2016-06-10 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics; Healthy non-elderly and elderly subjects; ASP2151; Safety
MeSH Terms: interventions — ASP2151

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- ASP2151 Low dose in non-elderly subjects group (Experimental): Subjects will receive ASP2151 daily on Days 1 to 7.
  Interventions: Drug: ASP2151
- ASP2151 High dose in non-elderly subjects group (Experimental): Subjects will receive ASP2151 daily on Days 1 to 7.
  Interventions: Drug: ASP2151
- ASP2151 Low dose in elderly subjects group (Experimental): Subjects will receive ASP2151 daily on Days 1 to 7.
  Interventions: Drug: ASP2151
- ASP2151 High dose in elderly subjects group (Experimental): Subjects will receive ASP2151 daily on Days 1 to 7.
  Interventions: Drug: ASP2151
- Placebo in non-elderly subjects group (Placebo Comparator): Subjects will receive matching placebo daily on Days 1 to 7.
  Interventions: Drug: Placebo
- Placebo in elderly subjects group (Placebo Comparator): Subjects will receive matching placebo daily on Days 1 to 7.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP2151 — Oral
  Arms: ASP2151 High dose in elderly subjects group; ASP2151 High dose in non-elderly subjects group; ASP2151 Low dose in elderly subjects group; ASP2151 Low dose in non-elderly subjects group
Drug: Placebo — Oral
  Arms: Placebo in elderly subjects group; Placebo in non-elderly subjects group

SUMMARY:
The objective of this study is to evaluate the safety and the pharmacokinetics of ASP2151 after multiple oral dosing of ASP2151 in healthy non-elderly male and elderly male Japanese subjects, and to compare the pharmacokinetics of ASP2151 in healthy non-elderly male and elderly male Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight: ≥50.0 kg and <85.0 kg
* Body mass index (BMI): ≥17.6 and <26.4 kg/m2

Exclusion Criteria:

* Subjects with a complication of any diseases
* Subjects with a history of hepatic disease
* Subjects with a history of heart disease
* Subjects with a history of respiratory disease
* Subjects with a history of alimentary disease
* Subjects with a history of renal disease
* Subjects with a history of cerebrovascular disorder
* Subjects with a history of malignant tumor
* Subjects with a history of drug allergies or allergies disorders excluding pollinosis
* Subjects with a history of drug dependency or alcohol dependence syndrome
* Subjects who developed genital herpes or herpes zoster within 90 days before the initial dosing
* Subjects who do not meet any of the criteria for laboratory tests
* Subjects who received medications within 14 days before the initial dosing.
* Subjects who received any investigational drugs in other clinical trials or post-marketing studies within 120 days before screening or the initial dosing
* Excessive alcohol drinking or smoking habit
* Subjects who previously received administration of ASP2151 (including placebo)
* Abnormalities detected on an ophthalmological examination
* Subjects who deviate from the normal range of standard 12-lead ECG at screening

Ages: 20 Years to 79 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-07; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of ASP2151 in plasma: Cmax | Up to Day 9
  Cmax: Maximum concentration
Pharmacokinetics of ASP2151 in plasma: tmax | Up to Day 9
  tmax: The time after dosing when Cmax occurs
Pharmacokinetics of ASP2151 in plasma: t1/2 | Up to Day 9
  t1/2: Apparent terminal elimination half-life
Pharmacokinetics of ASP2151 in plasma: C24 | Up to Day 9
  C24: Concentration at 24hours after dosing
Pharmacokinetics of ASP2151 in plasma: AUC24 | Up to Day 9
  AUC24: Area under the concentration-time curve from the time of dosing to 24hours after dosing
Pharmacokinetics of ASP2151 in plasma: AUCinf | Up to Day 9
  AUCinf: Area under the concentration-time curve from the time of dosing extrapolated to time infinity
Pharmacokinetics of ASP2151 in plasma: CL/F | Up to Day 9
  CL/F: Apparent total systemic clearance
Pharmacokinetics of ASP2151 in urine: Ae | Up to Day 9
  Ae: Amount excreted in urine
Pharmacokinetics of ASP2151 in urine: Cumulative Ae | Up to Day 9
Pharmacokinetics of ASP2151 in urine: Ae% | Up to Day 9
  Ae%: Percent of ASP2151 amount excreted in urine
Pharmacokinetics of ASP2151 in urine: Cumulative Ae% | Up to Day 9
Pharmacokinetics of ASP2151 in urine: CLR | Up to Day 9
  CLR: Renal clearance
Safety assessed by laboratory test: Hematology | Up to Day 14
Safety assessed by laboratory test: blood biochemistry | Up to Day 14
Safety assessed by laboratory test: urinalysis | Up to Day 14
Safety assessed by Vital sign measurement: axillary body temperature | Up to Day 14
Safety assessed by vital sign measurement: supine blood pressure | Up to Day 14
Safety assessed by vital sign measurement: supine pulse rate | Up to Day 14
Safety assessed by Standard 12-lead electrocardiogram | Up to Day 14
Safety assessed by Standard 12-lead electrocardiogram for QT assessment | Up to Day 14
Safety assessed by ophthalmological examination | Up to Day 14
Safety assessed by incidence of adverse events | Up to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Site JP00001, Osaka, Osaka, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kusawake T, Keirns JJ, Kowalski D, den Adel M, Groenendaal-van de Meent D, Takada A, Ohtsu Y, Katashima M. Pharmacokinetics and Safety of Amenamevir in Healthy Subjects: Analysis of Four Randomized Phase 1 Studies. Adv Ther. 2017 Dec;34(12):2625-2637. doi: 10.1007/s12325-017-0642-4. Epub 2017 Nov 13. PMID 29134426